CLINICAL TRIAL: NCT04669600
Title: A Multicenter, Phase 2a, Open-label, Non-randomized Study Evaluating the Efficacy, Safety, and Tolerability of BIVV020 in Adults With Persistent/Chronic Immune Thrombocytopenia (ITP)
Brief Title: A Phase 2a Study Evaluating BIVV020 in Adults With Persistent/Chronic Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDY16894; 2020-004162-18 (EudraCT Number); U1111-1253-2343 (Other: UTN)
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR445088 (Experimental): Participants received SAR445088 (BIVV020).
  Interventions: Drug: SAR445088 (BIVV020)

INTERVENTIONS:
Drug: SAR445088 (BIVV020) — Pharmaceutical form:solution for injection

SUMMARY:
Primary Objective:

- To evaluate the effect of BIVV020 on the durability of platelet response in participants with persistent/chronic immune thrombocytopenia (ITP)

Secondary Objectives:

* To assess the safety and tolerability of BIVV020
* To assess the pharmacokinetics of BIVV020
* To assess the response rate of treatment with BIVV020
* To assess the time to response
* To assess the effect of treatment with BIVV020 on the requirement for rescue ITP therapy
* To assess the immunogenicity of BIVV020

DETAILED DESCRIPTION:
Study duration:

* Screening period: up to 56 days
* Transition period between last sutimlimab dose and first dose of BIVV020 (for participants who were previously receiving sutimlimab): 14 days, included as part of the 56-day Screening period. Treatment duration: Minimum 52 weeks.

Visit frequency:

* Day 1
* Day 4
* Weeks 1 to 6: Weekly
* Weeks 7 to 12: Every other week
* Weeks 13 to 24: Every 4 weeks
* Weeks 25+: At least every 8 weeks
* End of Study visit: 22 weeks after the last dose of BIVV020

ELIGIBILITY:
Inclusion criteria :

* Male and female participants ≥18 years of age at the time of signing the informed consent
* Confirmed diagnosis of primary ITP; for participants who previously received sutimlimab in study TDR16218 (NCT03275454), a response to sutimlimab must have been obtained, as defined by platelet count ≥30 × 10^9/L on 2 visits at least 7 days apart
* For participants who have not previously received sutimlimab: persistent/chronic ITP (ITP lasting for ≥6 months) and all the following conditions:

  1. Platelet count ≤30 × 10^9/L on 2 occasions at least 5 days apart during the Screening Period;
  2. Lack of an adequate platelet count response (as defined by maintenance of sustained platelet count ≥30 × 109/L in the absence of bleeding) to at least 2 ITP treatments, 1 of which was a thrombopoietin receptor agonist. Other ITP treatments include: IVIg, anti-D immunoglobulin, corticosteroids, splenectomy, rituximab, cyclophosphamide, azathioprine, danazol, cyclosporin A, mycophenolate mofetil, or fostamatinib.
  3. If receiving weekly thrombopoietin receptor agonist dosing, the last dose must have been administered ≥7 days before the first dose of BIVV020. If receiving daily thrombopoietin receptor agonist dosing, the last dose must have been administered ≥24 hours before the first dose of BIVV020
  4. If applicable, concurrent administration of ITP medications (eg. corticosteroids, IVIg, azathioprine, danazol, cyclosporin A, mycophenolate mofetil, or thrombopoietin receptor agonists) is acceptable provided the participant has been on a stable dose for at least 1 month.
  5. If previously dosed with rituximab, the last dose of rituximab must have been administered at least 12 weeks before the first dose of BIVV020
* Documented vaccinations against encapsulated bacterial pathogens (Neisseria meningitidis, including serogroup B where available, Haemophilus influenzae, and Streptococcus pneumoniae) within 5 years of enrollment
* Contraceptive use for women of childbearing potential and men who were sexually active with a female partner of childbearing potential

Exclusion criteria:

Participants were excluded from the study if any of the following criteria apply:

* Clinically significant medical history or ongoing chronic illness that would jeopardize the safety of the participant or compromise the quality of the data derived from his/her participation in the study
* Clinical diagnosis of SLE
* Clinically relevant infection within the month prior to enrollment
* History of venous or arterial thrombosis within the year prior to enrollment
* Secondary ITP from any cause including lymphoma, chronic lymphocytic leukemia, and drug-induced thrombocytopenia
* Positive hepatitis B surface antigen (HBsAg) or active HCV infection
* HIV infection
* Pregnant or lactating women
* Hemoglobin level <10 g/dL

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (9):
- United States (2):
  - Investigational Site Number :8400001, Washington D.C., District of Columbia
  - Investigational Site Number :8400002, Tamarac, Florida
- Investigational Site Number :2030002, Ostrava - Poruba, Czechia
- Investigational Site Number :2760001, Essen, Germany
- Investigational Site Number :5280001, Leiden, Netherlands
- Spain (3):
  - Investigational Site Number :7240002, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number :7240001, Palma de Mallorca
  - Investigational Site Number :7240003, Seville
- Investigational Site Number :8260002, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PDY16894 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25319&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 centers in 5 countries. A total of 20 participants were screened from 04 Feb 2021 to 07 Sep 2021, of which 8 were screen failures due to not meeting eligibility criteria.
Pre-assignment Details: The study consisted of a screening period (up to 56 days), treatment period (up to 81 weeks), and follow-up visits (up to 22 weeks). A total of 12 participants [either switchers: who had received and responded to sutimlimab (BIVV009) in study TDR16218 (NCT03275454) or naïve: who have not previously received sutimlimab] were enrolled in this study.
Groups:
- SAR445088: Participants received a loading dose of SAR445088 (BIVV020) 50 milligram per kilogram (mg/kg) intravenously (IV) on Day 1, followed by maintenance doses of 600 mg subcutaneous (SC) weekly starting on Day 8 until the last participant enrolled completed 52 weeks of treatment. The maximum duration of treatment for an individual participant was up to 81 weeks.
Period: Overall Study
Arm/Group | SAR445088
Started | 12
Completed | 5
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Enrolled population consisted of all participants from screened population who had been allocated to a treatment regardless of whether the treatment was received or not.
Groups:
- SAR445088: Participants received a loading dose of SAR445088 (BIVV020) at 50 mg/kg IV on Day 1, followed by maintenance doses of 600 mg SC weekly starting on Day 8 until the last participant enrolled completed 52 weeks of treatment. The maximum duration of treatment for an individual participant was up to 81 weeks.
Arm/Group | SAR445088
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Durable Platelet Response
Description: A naive participant was a participant who did not use sutimlimab prior to enrollment. A switcher was a participant who used sutimlimab prior to enrollment. A naive participant was a responder if the platelet count was >=50 × 10^9/liter (L) at >=50 percent (%) of scheduled visits, or for participants with baseline platelet count <15 × 10^9/L, a >=20 × 10^9/L increase in platelet count from baseline at >=50% of scheduled visits, without receiving rescue immune thrombocytopenia (ITP) therapy. A switcher was a responder if the maintenance platelet count was >=30 × 10^9/L at >=50% of scheduled visits, without receiving rescue ITP therapy.
Time Frame: From Week 3 to Week 24
Population: Results are based on the overall number of participants analyzed = intent-to-treat (ITT) population which consisted of all exposed participants. Number analyzed = number of participants for each category (naive participant and switcher).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SAR445088
Number analyzed (Participants) | 12
percentage of participants
  Naive participant: number analyzed (Participants) | 8
  Naive participant | 0 [0.0 to 36.9]
  Switcher: number analyzed (Participants) | 4
  Switcher | 25 [19.4 to 99.4]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious AEs (SAE)
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. SAEs were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were AEs that developed after the first study treatment administration in the safety analysis period which was defined as the period from the first study intervention administration to the end of study (EOS) visit (up to Week 103).
Time Frame: From first study treatment administration (Day 1) up to Week 103
Population: The Safety population consisted of all enrolled participants who took at least 1 dose (including partial dose) of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR445088
Number analyzed (Participants) | 12
Participants
  Any TEAE | 8
  Any Treatment Emergent SAE | 2

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Hematology
Description: Criteria for potentially clinically significant laboratory abnormalities (PCSA): White blood cells: less than (<)3.0 Giga/L (Non-Black [NB]) or <2.0 Giga/L (Black [B]), greater than or equal to (>=)16.0 Giga/L; Lymphocytes: greater than (>)4.0 Giga/L; Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B); Monocytes: >0.7 Giga/L; Basophils: >0.1 Giga/L; Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN >=0.5 Giga/L); Hemoglobin: less than or equal to (<=) 115 grams per liter (g/L) (Male[M]) or <=95 g/L (Female[F]), >=185 g/L (M) or >=165 g/L (F), Decrease from baseline (DFB) >=20 g/L; Hematocrit: <=0.37 volume/volume (v/v) (M) or <=0.32 v/v (F); Red blood cells (RBC): >=6 Tera/L; Platelets:<100 Giga/L, >=700 Giga/L. Only the worst case during the treatment-emergent (TE) period for each participant with worsening from baseline is presented.
Time Frame: On Days 1, 15, 29, at Weeks 8, 12, 24, and then every 8 weeks until the end of study (EOS) (Week 103)
Population: Overall number of participants analyzed = safety population. Number analyzed = number of participants in the 'safety population' with available data for the corresponding categories. The Safety population consisted of all enrolled participants who took at least 1 dose (including partial dose) of study treatment. Only those participants with data available were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR445088
Number analyzed (Participants) | 12
Participants
  White blood cells: <3.0 Giga/L (NB) or <2.0 Giga/L (B) | 0
  White blood cells: >=16.0 Giga/L | 3
  Lymphocytes: >4.0 Giga/L | 2
  Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B): number analyzed (Participants) | 11
  Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B) | 0
  Monocytes: >0.7 Giga/L | 7
  Basophils: >0.1 Giga/L | 3
  Eosinophils: >0.5 Giga/L or >ULN (if ULN >=0.5 Giga/L) | 1
  Hemoglobin: <=115 g/L (M) or <=95 g/L (F) | 0
  Hemoglobin: >=185 g/L (M) or >=165 g/L (F) | 0
  Hemoglobin: DFB >=20 g/L | 0
  Hematocrit: <=0.37 v/v (M) or <=0.32 v/v (F) | 0
  RBC: >=6 Tera/L | 0
  Platelets: <100 Giga/L | 11
  Platelets: >=700 Giga/L | 0

4. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Clinical Chemistry
Description: Criteria for PCSA: Blood Urea Nitrogen: >=17 millimole (mmol)/L; Creatinine: >=150 micromole (mcmol)/L (Adults), >=30% and <100% change from baseline, >=100% change from baseline; Potassium: <3 mmol/L, >=5.5 mmol/L; Sodium: <=129 mmol/L, >=160 mmol/L; Aspartate Aminotransferase (AST): >3 ULN, >5 ULN, >10 ULN, >20 ULN; Alanine Aminotransferase (ALT): >3 ULN, >5 ULN, >10 ULN, >20 ULN; Alkaline Phosphatase (ALP): >1.5 ULN; Bilirubin: >1.5 ULN, >2 ULN; ALT and Total Bilirubin: ALT >3 ULN and TBILI >2 ULN. Only the worst case during the TE period for each participant with worsening from baseline is presented.
Time Frame: On Days 1, 15, 29, Weeks 8, 12 and 24, then every 8 weeks until the EOS (Week 103)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SAR445088
Number analyzed (Participants) | 12
Participants
  Blood Urea Nitrogen: >=17 mmol/L | 0
  Creatinine: >=150 mcmol/L (Adults) | 1
  Creatinine: >=30% and < 100% from baseline | 4
  Creatinine:>=100% from baseline | 1
  Potassium: <3 mmol/L | 0
  Potassium: >=5.5 mmol/L | 1
  Sodium:<=129 mmol/L | 0
  Sodium: >=160 mmol/L | 0
  AST: >3 ULN | 0
  AST: >5 ULN | 0
  AST: >10 ULN | 0
  AST: >20 ULN | 0
  ALT: >3 ULN | 0
  ALT: >5 ULN | 0
  ALT: >10 ULN | 0
  ALT: >20 ULN | 0
  ALP: > 1.5 ULN | 1
  Bilirubin: >1.5 ULN | 0
  Bilirubin: >2 ULN | 0
  ALT and total bilirubin: ALT>3ULN and TBILI >2ULN | 0

5. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Coagulation
Description: The number of participants with PCSA for coagulation parameters during the TE period without PCSA definition by biological function are presented. The parameters evaluated were prothrombin time, prothrombin international normalized ratio and activated partial thromboplastin time (APTT).
Time Frame: On Days 1, 15, 29, Weeks 8, 12 and 24, then every 8 weeks until the EOS (Week 103)
Population: Overall number of participants analyzed = Number of participants in the 'safety population' with available data for this outcome measure. Number analyzed = number of participants in the 'safety population' with available data for the corresponding categories. Some participants in 'Number Analyzed' were common for 2 or for all the 3 categories (Prothrombin time, Prothrombin International Normalized Ratio and APTT).
Measure: Count of Participants; unit: Participants
Arm/Group | SAR445088
Number analyzed (Participants) | 6
Participants
  Prothrombin time: <Lower limit of normal (LLN): number analyzed (Participants) | 3
  Prothrombin time: <Lower limit of normal (LLN) | 1
  Prothrombin time: >ULN: number analyzed (Participants) | 3
  Prothrombin time: >ULN | 2
  Prothrombin International Normalized Ratio: <LLN: number analyzed (Participants) | 4
  Prothrombin International Normalized Ratio: <LLN | 2
  Prothrombin International Normalized Ratio: >ULN: number analyzed (Participants) | 4
  Prothrombin International Normalized Ratio: >ULN | 2
  APTT: <LLN: number analyzed (Participants) | 4
  APTT: <LLN | 1
  APTT: >ULN: number analyzed (Participants) | 4
  APTT: >ULN | 3

6. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Urinalysis
Description: Criteria for PCSA: potential of Hydrogen (pH) <=4.6, >=8. Only the worst case during the TE period for each participant with worsening from baseline is presented.
Time Frame: On Days 1, 15, 29, Weeks 8, 12 and 24, then every 8 weeks until the EOS (Week 103)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SAR445088
Number analyzed (Participants) | 12
Participants
  pH: <=4.6 | 0
  pH: >=8 | 1

7. Secondary Outcome: Plasma Concentrations of SAR445088 (BIVV020)
Description: Plasma samples were collected at specified timepoints.
Time Frame: 1-hour post-dose on Day 1, on Days 8, 15, 29, 43, at Weeks 12, 16, 24, 32, 40, 48, 56, 64, 72, 80 and EOS visit, up to 103 weeks
Population: The Pharmacokinetic (PK) population consisted of all enrolled and treated participants (safety population) with at least 1 post-baseline PK sample. Only those participants with data available were included in the analysis.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | SAR445088
Number analyzed (Participants) | 12
microgram/milliliter (mcg/mL)
  Day 1: 1-hour post-dose | 1186.00 (254.24)
  Day 8: number analyzed (Participants) | 11
  Day 8 | 668.09 (139.19)
  Day 15: number analyzed (Participants) | 11
  Day 15 | 657.64 (107.33)
  Day 29: number analyzed (Participants) | 10
  Day 29 | 631.80 (64.52)
  Day 43: number analyzed (Participants) | 9
  Day 43 | 627.56 (84.39)
  Week 12: number analyzed (Participants) | 9
  Week 12 | 736.78 (164.07)
  Week 16: number analyzed (Participants) | 1
  Week 16 | 786.00 (NA) — Standard deviation could not be derived for a single participant.
  Week 24: number analyzed (Participants) | 8
  Week 24 | 781.63 (276.73)
  Week 32: number analyzed (Participants) | 6
  Week 32 | 695.67 (343.75)
  Week 40: number analyzed (Participants) | 6
  Week 40 | 602.33 (385.64)
  Week 48: number analyzed (Participants) | 6
  Week 48 | 559.33 (300.73)
  Week 56: number analyzed (Participants) | 5
  Week 56 | 602.80 (224.08)
  Week 64: number analyzed (Participants) | 5
  Week 64 | 615.80 (247.91)
  Week 72: number analyzed (Participants) | 4
  Week 72 | 584.25 (243.37)
  Week 80: number analyzed (Participants) | 2
  Week 80 | 602.50 (287.79)
  EOS (Week 103): number analyzed (Participants) | 10
  EOS (Week 103) | 206.46 (157.42)

8. Secondary Outcome: Number of Responders to SAR445088 (BIVV020)
Description: A participant was a responder if the platelet count was >=50 × 10^9/L and there was a greater than 2-fold increase from baseline, measured on 2 occasions at least 7 days apart with the absence of bleeding [bleeding score >=2 on the World Health Organization (WHO) bleeding scale] while the platelet counts were maintained above the threshold and lack of combination ITP therapy during this period. WHO bleeding scores: 1=Petechiae; 2=Mild blood loss; 3=Gross blood loss; and 4=Debilitating blood loss.
Time Frame: At Weeks 24 and 56
Population: The ITT population consisted of all exposed participants.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR445088
Number analyzed (Participants) | 12
Participants
  Week 24 | 2
  Week 56 | 2

9. Secondary Outcome: Time to First Platelet Response
Description: Time to first platelet response was defined as greater than or equal to each of the following values: 50 × 10^9/L or 100 × 10^9/L (confirmed by 2 measurements at least 7 days apart). It was calculated as date of first occurrence of confirmed platelet count response before rescue therapy.
Time Frame: From Baseline (Day 1) up to Week 56
Population: Overall number of participants analyzed = ITT Population which consisted of all exposed participants. Number analyzed = number of participants in the 'ITT Population' who met the specified platelet counts (>=50 x10^9/L or >=100 x10^9/L) as confirmed by 2 measurements at least 7 days apart. Participants who met the criteria 'Platelet count >=100 x10^9/L' were the same as who met the criteria 'Platelet count >=50 x10^9/L'.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | SAR445088
Number analyzed (Participants) | 12
weeks
  Platelet count>=50 x 10^9/L: number analyzed (Participants) | 4
  Platelet count>=50 x 10^9/L | 18.5 [13.5 to 49.5]
  Platelet count>=100 x 10^9/L: number analyzed (Participants) | 4
  Platelet count>=100 x 10^9/L | 18.5 [13.5 to 49.5]

10. Secondary Outcome: Percentage of Participants Who Did Not Require Rescue Therapy for an Acute Episode of Thrombocytopenia After Week 3
Description: Data was collected to assess the effect of treatment with SAR445088 (BIVV020) on the requirement for rescue ITP therapy.
Time Frame: Up to Week 84
Population: The ITT population consisted of all exposed participants.
Measure: Number; unit: percentage of participants
Arm/Group | SAR445088
Number analyzed (Participants) | 12
percentage of participants
  Week 3 to Week 24 during treatment period | 75.0
  Week 3 to Week 56 during treatment period | 75.0
  Week 3 to the end of on-treatment period | 75.0

11. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADAs) Response to SAR445088 (BIVV020)
Description: Plasma samples were analyzed for the presence of ADAs for SAR445088 (BIVV020) using validated assays. Treatment-induced ADA was defined as ADAs that developed during the treatment-emergent period and without pre-existing ADA. Pre-existing ADA was defined as ADAs present in samples drawn before first study treatment administration. Treatment-boosted ADA positive was defined as pre-existing ADA (i.e., ADA positive at baseline) that was boosted at least a 9-fold increase of titer values during the treatment-emergent period than the baseline. Treatment-emergent ADA positive was defined as either treatment-induced ADA positive or treatment-boosted ADA positive during the treatment-emergent period. Inconclusive ADA was defined as the one that could not irrefutably be classified as with or without treatment-emergent ADA.
Time Frame: Up to Week 103
Population: The ADA population consisted of all enrolled and treated participants (safety population) with at least 1 post-baseline ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR445088
Number analyzed (Participants) | 12
Participants
  Participants with ADA negative or missing at baseline | 11
  Participants with treatment-induced ADA | 0
  Participants with pre-existing ADA | 1
  Participants with treatment-boosted ADA | 0
  Participants with treatment-emergent ADA during 24-week treatment period | 0
  Participants with treatment-emergent ADA during 52-week treatment period | 0
  Participants without treatment-emergent ADA | 12
  Participants with inconclusive ADA | 0

ADVERSE EVENTS:
Time Frame: The TEAEs were collected from first study treatment administration (Day 1) up to Week 103
Description: The Safety population consisted of all enrolled participants who took at least 1 dose (including partial dose) of study treatment. As prespecified, AEs recorded for doses 50 mg/kg (loading dose) and 600 mg (maintenance dose) of SAR445088 are presented under the reporting group, SAR445088.
Arm/Group | SAR445088
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR445088 (N=12)
Appendicitis (Infections and infestations) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR445088 (N=12)
Covid-19 (Infections and infestations) | 3 (4)
Influenza (Infections and infestations) | 1 (2)
Post-Acute Covid-19 Syndrome (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Burning Sensation (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Eye Irritation (Eye disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Injection Site Bruising (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Blood Cholesterol Increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT04669600/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT04669600/SAP_001.pdf